CLINICAL TRIAL: NCT06205160
Title: The EpiGrid Study Evaluation of New Flexible High-density Intra-operative ECoG Electrodes for Epilepsy Surgery
Brief Title: Evaluation of New Flexible High-density Intra-operative ECoG Electrodes for Epilepsy Surgery. ( EpiGrid )
Acronym: EpiGrid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurosoft Bioelectronics SA (Industry)
Collaborators: UMC Utrecht (Other); European Research Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-01202
Record Dates: First submitted 2023-12-19; First posted 2024-01-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Focal Epilepsy; Intraoperative Monitoring
Keywords: intra-operative electrocorticography; HFO; epileptic biomarkers; high frequency oscillations; epilepsy surgery; flexible ECoG; subdural electrode
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental)
  Interventions: Device: SOFT ECoG subdural grid electrode

INTERVENTIONS:
Device: SOFT ECoG subdural grid electrode — Test Device (SOFT ECoG subdural grid electrode): used for recording. During epilepsy surgery, in addition to standard clinical protocol (recording with comparator device), subjects will undergo ≥ 2 additional intracranial recordings with the SOFT ECoG flexible high density electrode grid (TD). Recording will be registered pre- and post-resection.
  All procedures will be conducted according to standard clinical practice. Any medical decision making will be done using the standard of care CE-marked device (CD). The investigational, non-CE marked device is not used for clinical decision making.

SUMMARY:
The objective of this prospective interventional monocentric clinical investigation is to evaluate the feasibility and performance of the flexible high-density SOFT ECoG electrode grids, manufactured by Neurosoft Bioelectronics SA (test device; TD), in comparison to regular high-density electrode grids (ADTech, CE-marked) (control device; CD) routinely used at the investigation site during epilepsy surgery.

Subjects will undergo ≥ 2 additional intracranial recordings pre- and post-resection with the TD next to the standard recordings with the CD during ECoG-tailored epilepsy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of enrolment
* Lesional epilepsy (incl. secondary mesial temporal sclerosis) that is considered a candidate for intra-operative high-density grid recordings (incl. patients who underwent sEEG preceding resective surgery)
* Provided informed consent for study participation by the subject

Exclusion Criteria:

* Occipital lesion
* Surgeries involving a primary mesial temporal lesion, a disconnection, or hemispherectomy.
* Planned ioECoG recordings during fully awake surgery and/or functional recordings
* Use of anticoagulants that cannot be discontinued during the perioperative period, or a factor XIII deficiency or any other haematological disease
* Active participation in another investigational device study
* Any other condition that in the opinion of the investigator may adversely affect the safety of the subject or would limit the subject's ability to complete the study.
* Insufficient understanding of Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Background SNR pre-resection recording | up to 24 hours
  Performance in terms of signal quality is assessed via background signal to noise ratio (SNR). Only channels which record properly based on visual inspection (no noise, no flat line) will be included in the background SNR calculation. For the pre-resection recordings (SITUATION I/I*), the background SNR per (included) channel and the average SNR for the electrode grid will be calculated, and pairwise comparison will be conducted between TD (SITUATION I*) and CD (SITUATION I).

SECONDARY OUTCOMES:
Electrode deficiency ratio (%) | up to 24 hours
  The individual electrodes will be classified, per recording, as poor or good signal quality based on visual criteria (i.e., noise, flat signal due to overlap with resection cavity or silicone of secondary electrode strip, pulsation artifacts). As a result, an electrode deficiency ratio (%) will be calculated as follows: # bad electrodes divided by the total # of electrodes per recording. This will be determined for the similar positioned CD recording (SITUATION I/II) to allow comparison with the TD (SITUATION I*/I**).
Epileptic biomarker identification ( eg. number of spikes/HFOs per min, event SNR) | up to 24 hours
  After the surgery, spikes and high frequency oscilations (HFOs) will be visually marked in the final minute of the recording (note: assisted by automated spike/HFO detector) and checked by an expert. Marking of spikes and HFOs will be done in the TD and the corresponding CD recordings pre- and post-resection. Event rates (number of spikes/HFOs per minute) per channel and total per recording will be compared between the TD and CD. The average event SNR per channel and the average SNR per epileptogenic event type will be calculated per recording. The event SNR will be compared between the CD recording (SITUATION I/II) and the TD (SITUATION I*/I**).
Background SNR of post-resection recordings | up to 24 hours
  The background SNR for post-resection recordings (SITUATION II/II**) will be computed and pairwise compared. Note that it shall be considered that for the post-resection recordings (SITUATION II/II**), in particular when measuring near/in the resection cavity, the performance of both the TD and CD for electrode deficiencies might differ significantly, positively and negatively.
Surgical complications (e.g. SAEs/SADEs) | up to hospital discharge, on average at 10 days
  The safety analysis will include surgical complications in terms of device deficiencies (DDs) and serious adverse events (SAEs), and whether these are device related (SADEs).
Usability evaluation | up to 48 hours
  A (digital) usability questionnaire (system usability scale + open questions) will be collected (within 48h after surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center (UMC) Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No